CLINICAL TRIAL: NCT02882100
Title: Adjuvanted Influenza Vaccination and Morbidity and Mortality in U.S. Nursing Homes
Brief Title: Adjuvanted Influenza Vaccination in U.S. Nursing Homes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insight Therapeutics, LLC (Other)
Collaborators: Case Western Reserve University (Other); Brown University (Other); Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INSI-201603
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Influenza; Influenza-like Illness
Keywords: influenza; vaccine; vaccination; nursing home; cluster randomized trial; respiratory-related hospitalization
MeSH Terms: conditions — Influenza, Human | interventions — fluad vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aTIV (Experimental): NH facilities randomized to receive adjuvanted trivalent influenza vaccine (aTIV, FLUAD) for the residents
  Interventions: Biological: adjuvanted trivalent influenza vaccine; Biological: trivalent influenza vaccine
- TIV (Active Comparator): NH facilities randomized to receive standard trivalent influenza vaccine (TIV, Fluvirin) for the residents
  Interventions: Biological: trivalent influenza vaccine

INTERVENTIONS:
Biological: adjuvanted trivalent influenza vaccine — Nursing home residents over 65 years are allocated to receive adjuvanted trivalent vaccine. Residents under 65 years are provided standard trivalent vaccine (TIV-Fluvirin).
  Other Names: Fluad; aTIV
  Arms: aTIV
Biological: trivalent influenza vaccine — Nursing home residents are allocated to receive standard trivalent vaccine (TIV).
  Other Names: Fluvirin; TIV

SUMMARY:
This study is powered to prospectively evaluate the relative effectiveness of adjuvanted trivalent influenza vaccine (aTIV; FLUAD) in preventing influenza mortality, hospitalization, and functional decline in a nursing home population in the U.S., compared to the commercially available, standard dose trivalent seasonal influenza vaccine (TIV; Fluvirin).

DETAILED DESCRIPTION:
SUMMARY: A random study sample of up to 1000 NHs within 75 miles of the local area of the 121 cities where the CDC performs weekly influenza surveillance (estimated N= 11,239) may be offered the opportunity for participation; the first 1000 eligible to participate and accepting the offer will be enrolled. Participating facilities will be offered vaccine education for residents and staff, but will be randomly allocated to receive aTIV (FLUAD) vaccine or usual care (TIV) vaccination for their residents.

BACKGROUND: Lower respiratory tract infection (LRI), including pneumonia, bronchitis, and tracheobronchitis, is the leading cause of infectious mortality and hospitalization in older adults , and nursing home (NH) residents. Pneumonia and infection often produce attenuated signs and symptoms in older adults, leading to delayed or even misdiagnosis for this population. Diagnosis is further compromised due to few and sporadic clinician visits with nursing home residents, and reduced access to radiology. LRI may or may not directly lead to hospitalization, but LRIs are associated with considerable other morbidity than can result in hospitalization, including exacerbation of underlying cardiopulmonary diseases. Hospitalization rates for NH residents vary considerably between facilities, but the majority of hospitalizations occur during the 12 weeks during which influenza peaks each year.

OBJECTIVES: The primary objective is to estimate the differences in hospitalization rates during influenza season experienced by long-stay nursing home residents, between facilities using adjuvanted trivalent vaccine vs. standard trivalent vaccine. The secondary objective is to estimate the differences in the likelihood of Activities of Daily Living (ADL) functional decline and mortality rates in the study nursing homes, and influenza outbreaks.

ELIGIBILITY:
Inclusion Criteria:

* Long-term care facilities within 75 miles of one of the 121 cities that serve as CDC surveillance sites

Exclusion Criteria:

* Facilities that used high dose influenza vaccine in residents over age 65 in previous influenza season (2015-16)
* Facilities having fewer than 50 long-stay residents
* Hospital-based facilities
* Facilities with more than 20% of the population under age 65
* Facilities not submitting Minimum Data Set (MDS) data

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 823 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Hospitalization for a respiratory-related Illness | up to 1 year
  Time to first occurrence of hospitalization for a respiratory-related Illness based upon Medicare inpatient hospital claims
Hospitalization for all causes | up to 1 year
  Time to first occurrence of hospitalization for all-causes

SECONDARY OUTCOMES:
Activities of daily living (ADL) scores | up to 1 year
  Change in activities of daily living (ADL) scores
Mortality | up to 1 year
  Difference in mortality rate

OTHER OUTCOMES:
Influenza outbreaks | up to 1 year
  Difference in occurrence of documented influenza outbreaks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gravenstein, MD, MPH, Principal Investigator — Case Western Reserve Univsity; Vincent Mor, PhD, Principal Investigator — Brown University; H. Edward Davidson, PharmD, MPH, Principal Investigator — Insight Therapeutics, LLC
Locations (1):
- Insight Therapeutics, LLC, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Bridges CB, Cox NJ, Fukuda K. Influenza-associated hospitalizations in the United States. JAMA. 2004 Sep 15;292(11):1333-40. doi: 10.1001/jama.292.11.1333. PMID 15367555
- [Background] Hayward AC, Harling R, Wetten S, Johnson AM, Munro S, Smedley J, Murad S, Watson JM. Effectiveness of an influenza vaccine programme for care home staff to prevent death, morbidity, and health service use among residents: cluster randomised controlled trial. BMJ. 2006 Dec 16;333(7581):1241. doi: 10.1136/bmj.39010.581354.55. Epub 2006 Dec 1. PMID 17142257
- [Derived] Smith CL, Bednarchik B, Aung H, Wilk DJ, Boxer RS, Daddato AE, Wilson BM, Gravenstein S, Canaday DH. Humoral and Cellular Immunity Induced by Adjuvanted and Standard Trivalent Influenza Vaccine in Older Nursing Home Residents. J Infect Dis. 2023 Sep 15;228(6):704-714. doi: 10.1093/infdis/jiad071. PMID 36951196
- [Derived] Gravenstein S, McConeghy KW, Saade E, Davidson HE, Canaday DH, Han L, Rudolph J, Joyce N, Dahabreh IJ, Mor V. Adjuvanted Influenza Vaccine and Influenza Outbreaks in US Nursing Homes: Results From a Pragmatic Cluster-Randomized Clinical Trial. Clin Infect Dis. 2021 Dec 6;73(11):e4229-e4236. doi: 10.1093/cid/ciaa1916. PMID 33400778
- [Derived] McConeghy KW, Davidson HE, Canaday DH, Han L, Saade E, Mor V, Gravenstein S. Cluster-randomized Trial of Adjuvanted Versus Nonadjuvanted Trivalent Influenza Vaccine in 823 US Nursing Homes. Clin Infect Dis. 2021 Dec 6;73(11):e4237-e4243. doi: 10.1093/cid/ciaa1233. PMID 32882710
- See also: FDA approves first seasonal influenza vaccine containing an adjuvant — https://wayback.archive-it.org/7993/20170111160747/http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm474295.htm